CLINICAL TRIAL: NCT02455687
Title: Two Doses of the Intravenous Magnesium Sulfate Versus the Standard Single Dose With/Without Nebulized Budesonide for the Emergency Management of the Severe Asthma. A Randomized Controlled Trial.
Brief Title: Two Doses of the Intravenous Magnesium Sulfate Versus the Standard Single Dose ,With/ Without the Nebulized Budesonide For the Management of the Severe Asthma Exacerbation in the Emergency Room; A Randomized Controlled Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1400046
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2023-12

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma; Intravenous magnesium sulfate; Inhaled budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Hi-Mg + Bud (Active Comparator): Group one will receive a high,then standard dose of intravenous magnesium sulfate with blinded nebulized budesonide.
  Interventions: Drug: Hi-dose iv MgSO4; Drug: Nebulized budesonide
- Hi-Mg + P (Placebo Comparator): Group two will receive a high,then standard dose of intravenous magnesium sulfate with blinded nebulized normal saline.
  Interventions: Drug: Hi-dose iv MgSO4; Drug: Nebulized normal saline
- Std-Mg + Bud (Active Comparator): Group three will receive a single standard dose of intravenous magnesium sulfate plus one dose of intravenous normal saline with blinded nebulized budesonide.
  Interventions: Drug: Nebulized budesonide; Drug: Std-dose iv MgSO4
- St-Mg + P (Placebo Comparator): Group four will receive a single dose of intravenous magnesium sulfate plus one dose of intravenous normal saline with blinded nebulized normal saline
  Interventions: Drug: Std-dose iv MgSO4; Drug: Nebulized normal saline

INTERVENTIONS:
Drug: Hi-dose iv MgSO4
  Arms: Hi-Mg + Bud; Hi-Mg + P
Drug: Nebulized budesonide
  Other Names: Pulmicort
  Arms: Hi-Mg + Bud; Std-Mg + Bud
Drug: Std-dose iv MgSO4
  Arms: St-Mg + P; Std-Mg + Bud
Drug: Nebulized normal saline
  Arms: Hi-Mg + P; St-Mg + P

SUMMARY:
Many studies have investigated the efficacy and safety of Intravenous magnesium sulfate and inhaled steroids in addition to the standard treatment for patients with severe asthma attacks.

In this 2x2 factorial design blinded randomized study, no interaction of hypothesized treatments is expected.Investigators hypothesize that two doses of intravenous magnesium sulfate,a high dose followed by a (lower) standard dose, will shorten the time to medical readiness for discharge compared to a single standard dose followed by placebo.The second hypothesis is that nebulized inhaled budesonide will be superior to placebo.

DETAILED DESCRIPTION:
Patient with a severe asthma attack will be admitted to the observation area in the Pediatric Emergency Center and assessed for eligibility for the study by the attending physician, based upon our study inclusion/exclusion criteria.

Eligible patients will be enrolled after obtaining written consent from the parents. Patients will receive routine treatment for a severe asthma attack, such as inhaled bronchodilators, plus intravenous steroids and supplementary oxygen if needed. Standard blood work and chest X-Ray will be obtained and bronchial asthma severity score will be measured at baseline before starting treatment,and then at 4,8,12,24,36,48 hr and thereafter. The medical team as well as parents and patient will be blinded to the medications delivered. The patient will be randomized into one of the four study groups and adverse effects of the medications in each group will be monitored and documented carefully.

ELIGIBILITY:
Inclusion Criteria:

1. Children 2-14 years of age.
2. Known to have bronchial asthma.
3. Presenting in severe asthma exacerbation
4. Asthma severity score 8 or higher according to PRAM asthma severity .

Exclusion Criteria:

1. Prematurity <34 weeks of gestation.
2. Critically ill children requiring immediate intubation or ICU admission.
3. Transfers from other institutions.
4. Adverse drug reaction or allergy to budesonide,salbutamol,ipratropium bromide, prednisone, prednisolone, methylprednisolone, or magnesium sulfate.
5. History of neuromuscular disease, cardiac disease, renal disease, liver disease.
6. Underlying chronic lung disease.
7. Radiographic evidence of pneumonia or lung collapse .
8. Hemodynamic instability.
9. Instrumented airway or Tracheotomy.
10. Colostomy or ileostomy.
11. Malabsorption disorder.
12. Known vitamin D deficiency.
13. Receiving Milk of Magnesium for Constipation
14. Chronic diarrhea (duration for 2 weeks)
15. Diuretics use.
16. Immunodeficiency.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Time to medical readiness for discharge. | 3 years
  The aim of the study is to find out if the two doses of intravenous magnesium sulfate 100 mg/kg followed by 50 mg/kg with or without nebulized budesonide would shorten the length of the emergency center's stay in comparison to the 50 mg/kg dose with or without nebulized budesonide in treating severe asthma attack in children, who are admitted to the pediatric emergency center Al-Sadd, in a double blinded randomized controlled trial. .

SECONDARY OUTCOMES:
Overall length of the hospital stay (hours/days) . | 3 years
  Would the two doses of intravenous magnesium sulfate with or without nebulized budesonide shorten the length of the emergency center's stay in treating severe asthma attack in children, compared to the 50 mg/kg dose with or without nebulized budesonide?
The rate of admission to pediatric intensive care unit (%) | 3 years
  Would the two doses of intravenous magnesium sulfate with or without nebulized budesonide decrease the PICU admission rate in treating severe asthma attack in children, compared to the 50 mg/kg dose with or without nebulized budesonide?
Comparison of clinical response in severity score (%) | 3 years
  Would the two doses of intravenous magnesium sulfate with or without nebulized budesonide decrease the asthma severity score at 4, 8,12,24,36,48,60,72 hours in treating severe asthma attack in children, compared to the 50 mg/kg dose with or without nebulized budesonide?
Frequency of need for revisit and readmission to pediatric emergency center for same diagnosis(%) | 3 years
  Would the two doses of intravenous magnesium sulfate with or without nebulized budesonide decrease revisit to emergency services in treating severe asthma attack in children, compared to the 50 mg/kg dose with or without nebulized budesonide?
  Would the two doses of intravenous magnesium sulfate with or without nebulized budesonide decrease readmission rate in treating severe asthma attack in children, compared to the 50 mg/kg dose with or without nebulized budesonide? •

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Alansari, MD, Study Director — Sidra Medicine
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided